CLINICAL TRIAL: NCT00320918
Title: Chart Review on Patients With Unresectable/Metastatic Cholangiocarcinoma Treated in the UNM Cancer Center With a Combination of Irinotecan, Capecitabine and Celecoxib
Brief Title: Chart Review: Unresectable/Metastatic Cholangiocarcinoma Treated With Irinotecan, Capecitabine and Celecoxib
Status: Terminated | Type: Observational
Why Stopped: This was a Chart Review only and was entered in the system in error.
Sponsor: University of New Mexico (Other)
Responsible Party: Fa-Chyi Lee, MD; Principal Investigator, University of New Mexico - CRTC
Other Study IDs: 4504C
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Cholangiocarcinoma
Keywords: Unresectable/metastatic cholangiocarcinoma; Cancer; Chart Review
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chart Review on Patients with unresectable/metastatic cholangiocarcinoma treated in the UNM Cancer Center with a combination of irinotecan, capecitabine and celecoxib.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable/metastatic cholangiocarcinoma treated in the UNM Cancer Center with a combination of irinotecan, capecitabine and celecoxib.

Exclusion Criteria:

* Not specified.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable/metastatic cholangiocarcinoma treated in the UNM Cancer Center with a combination of irinotecan, capecitabine and celecoxib.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States